CLINICAL TRIAL: NCT06603974
Title: An Exploratory Study of Benmelstobart in Combination with Antiangiogenesis Drugs and Neoadjuvant Chemotherapy for Locally Progressive Gastric Cancer / Gastroesophageal Junction Carcinoma
Brief Title: The Efficacy and Safety of Benmelstobart for GC/EGC
Acronym: EASOBFGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQXB-GC-001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative; Tegafur; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benmelstobart combined with antiangiogenic drugs and neoadjuvant chemotherapy (Experimental): Benmelstobart: 1200mg, diluted to 250ml with normal saline, infusion time 60 ± 10mins. The first day of each cycle, 3 weeks (21 days) as a treatment cycle; antiangiogenic drugs are decided by the investigator according to the actual situation; tegafur: it needs to be administered according to the patient's body surface area< 40mg / time at 1.25m2; > 50mg/ time for 1.25m2 and <1.5m2; > 60mg/ time at 1.5m2; Oral, twice a day, after morning and evening meals, for 14 consecutive days, rest for 7 days, as a treatment cycle; Repeat every 3 weeks; oxaliplatin: 130mg/m2, administered on the first day of each cycle, repeated every 3 weeks; Chemotherapy drugs can also be selected by the investigator.
  albumin paclitaxel: 260mg/m2, intravenous infusion, 30 minutes per infusion, once every 3 weeks, administered on the first and eighth days of each cycle
  Interventions: Procedure: surgery; Drug: Benmelstobart; Drug: tegafur; Drug: oxaliplatin; Drug: albumin paclitaxel

INTERVENTIONS:
Procedure: surgery — After receiving the corresponding neoadjuvant treatment for 2 cycles, surgery was performed within 3-6 weeks after drug withdrawal.
Drug: Benmelstobart — 1200mg, diluted to 250ml with normal saline, infusion time 60 ± 10mins. The first day of each cycle, 3 weeks (21 days) as a treatment cycle
Drug: tegafur — it needs to be administered according to the patient's body surface area< 40mg / time at 1.25m2; > 50mg/ time for 1.25m2 and <1.5m2; > 60mg/ time at 1.5m2; Oral, twice a day, after morning and evening meals, for 14 consecutive days, rest for 7 days, as a treatment cycle; Repeat every 3 weeks;
Drug: oxaliplatin — 130mg/m2, administered on the first day of each cycle, repeated every 3 weeks;
Drug: albumin paclitaxel — 260mg/m2, intravenous infusion, 30 minutes per infusion, once every 3 weeks, administered on the first and eighth days of each cycle

SUMMARY:
The goal of this clinical trial is to evaluate the major pathological response (MPR) rate of locally advanced gastric cancer / gastroesophageal junction cancer treated with bemosumab combined with antiangiogenic drugs and neoadjuvant chemotherapy.

Researchers will use drug Benmelstobart in combination with antiangiogenesis drugs and newadjuvant chemotherapy to see if the drug works to treat locally advanced gastric cancer / gastroesophageal junction cancer.

Participants will:injection drug Benmelstobart，On the first day of each cycle, 3 weeks (21 days) were a treatment cycle.

DETAILED DESCRIPTION:
The phase i/ii clinical study of benmelstobart combined with anlotinib, oxaliplatin and capecitabine in the first-line treatment of gastric / gastroesophageal junction adenocarcinoma has shown good efficacy and safety. Anti vascular drugs have also shown excellent anti-tumor effects in the neoadjuvant treatment of locally advanced gastric cancer. Therefore, this study plans to explore the efficacy of benmelstobart combined with anti angiogenic drugs and neoadjuvant chemotherapy for locally advanced gastric cancer / gastroesophageal junction cancer, and make up for this part of the treatment gap.

ELIGIBILITY:
Inclusion Criteria:

* 1.18 ≤ 70 years old, male or female;
* 2. ECoG score 0-1;
* 3. patients with locally advanced gastric cancer / gastroesophageal junction cancer confirmed by pathology (histology or cytology) (according to the WHO classification in 2015);
* 4. according to the eighth edition of clinical tumor TNM staging, patients with t3~4n+m0 gastric cancer / gastroesophageal junction cancer confirmed to be resectable or potentially resectable by endoscopic ultrasound and enhanced CT;
* 5. have measurable lesions (according to RECIST 1.1 standard, the long diameter of CT scan of tumor lesions is ≥ 10mm, and the short diameter of CT scan of lymph node lesions is ≥ 15mm;), and the tumor is > 2cm directly;
* 6. patients who were initially diagnosed with gastric cancer / gastroesophageal junction cancer without radiotherapy, chemotherapy, surgery and targeted therapy before enrollment;
* 7. if the main organ function is normal, it meets the following criteria:

  1. Blood routine examination must meet the following requirements (no blood transfusion, no use of hematopoietic factors and no use of drugs for correction within 14 days):

     1. ANC ≥ 1.5 × 109/l;
     2. PLT ≥ 100 × 109/l;
     3. HB ≥ 90 g/L；
  2. Biochemical tests must meet the following criteria:

     1. TBIL ≤ 1.5 × ULN;
     2. Alt, AST ≤ 2.5 × ULN
     3. Serum creatinine SCR ≤ 1.5 × ULN, endogenous creatinine clearance ≥ 50 ml / min (Cockcroft Gault formula);
  3. Coagulation function must meet: INR ≤ 1.5 × ULN and APTT ≤ 1.5 × ULN;
* 8. patients with grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 450ms (male), QTc ≥ 470ms (female)) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
* 9. female subjects of childbearing age must have a serum pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraceptive measure (such as IUD, contraceptive or condom) during the study period and within 3 months after the last administration of study medication; For male subjects whose partner is a female of childbearing age, they should be surgically sterilized, or agree to use effective methods of contraception during the study and within 3 months after the last study administration; The subjects voluntarily joined the study and signed the informed consent form. -10.The compliance was good and they cooperated with the follow-up;

Exclusion Criteria:

* 1. exclusion criteria of target disease

  1. Patients with distant metastasis;
  2. Subjects who had previously received anti-PD-1 (L1) or CTLA4 mAb therapy;
* 2. medical history and comorbidities

  1. Other malignant tumors in the past 3 years;
  2. Have any history of active autoimmune disease or autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy)); Patients with vitiligo or childhood asthma have been completely relieved and can be included without any intervention in adults; Patients who needed bronchodilators for medical intervention could not be included;
  3. Immunosuppressive drugs used within 14 days before the first use of study drugs, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (i.e. no more than 10 mg/ day prednisone or its equivalent);
  4. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg despite optimal medical treatment);
  5. Patients with newly diagnosed angina within 3 months before screening or myocardial infarction within 6 months before screening; Arrhythmias (including QTCF: ≥ 450 ms for men and ≥ 470 MS for women) require long-term use of antiarrhythmic drugs and New York Heart Association class ≥ II cardiac insufficiency; Or uncontrollable heart failure;
  6. There is evidence that there are previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiologic pneumonia, drug-induced pneumonia and severe impairment of lung function;
  7. Complicated with severe infection within 4 weeks before the first administration (such as requiring intravenous infusion of antibiotics, antifungal or antiviral drugs), or fever of unknown cause >38.5 ° C during the screening period / before the first administration;
  8. Clinically significant hemoptysis (more than 50 ml hemoptysis per day) within 3 months before the study, or clinically significant bleeding symptoms or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood + + or above the baseline, or suffering from vasculitis, etc.).
  9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
  10. Live attenuated vaccine was administered within 4 weeks before the first dose or planned during the study;
* 3. physical examination and laboratory examination

  1. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 iu/ml), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analysis method), or combined hepatitis B and C co infection;
  2. Pregnant or lactating women; Patients with fertility are unwilling or unable to take effective contraceptive measures;
  3. Known to have a positive history of human immunodeficiency virus (HIV) examination or known to have acquired immune deficiency syndrome (AIDS);
* 4. allergy, anaphylaxis and adverse drug reactions

  1. Severe allergic reaction to other monoclonal antibodies;
  2. Allergy or intolerance to infusion;
  3. Have a history of severe allergy to antiangiogenic drugs or their preventive drugs;
* 5. subjects who are participating in other clinical studies or whose first medication time is less than 4 weeks from the end of the previous clinical study (the last medication), or who have 5 half lives of the study drug;
* 6. the subject is known to have a history of psychotropic substance abuse, alcohol abuse or drug abuse;
* 7. the investigator believes that there are any conditions that may damage the subject or cause the subject to be unable to meet or perform the research requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-16 (Estimated); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 2 years
  Tumor tissue samples surgically removed after neoadjuvant therapy, without residual tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, master, Study Chair — Department of Digestive Surgery, Xijing Hospital, Air Force Medical University